CLINICAL TRIAL: NCT06649136
Title: An International, Multicentre, Interventional, Randomised, Assessor-blinded Trial to MAXimise the METHotrexate Therapy Potential in Patients with Active Rheumatoid Arthritis
Brief Title: MethMax Trial: MAXimising the METHotrexate Therapy Potential in Patients with Active Rheumatoid Arthritis
Acronym: MethMax
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Leiden University Medical Center (Other); Karolinska Institutet (Other); Queen Mary University of London (Other); Diakonhjemmet Hospital AS (Unknown)
Responsible Party: Principal Investigator, Helga Lechner-Radner, Medical University of Vienna, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MethMax Trial
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; methotrexate; therapy adherence; biomarker
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: joint assessor blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methotrexate 25mg s.c. (Active Comparator): methotrexate 25mg s.c. weekly dose
  Interventions: Drug: Methotrexate
- methotrexate 25mg p.o. (Active Comparator): methotrexate 25mg p.o. weekly dose
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — comparison between oral and subcutaneous methotrexate dosis of 25mg

SUMMARY:
The MethMax trial is a prospective, international, multicentre, randomised, assessor-blinded, parallel-group, low intervention study. Patients with active rheumatoid arthritis treated with oral methotrexate up to 25mg weekly will be randomised in 50:50 fashion to receive 25mg oral vs subcutaneous methotrexate for the period of 24 weeks. In regular visits, patient reported outcomes, clinical disease activity, therapy adherence and diverse established and exploratory biomarkers will be assessed.

DETAILED DESCRIPTION:
Methotrexate is recommended as the first-line therapy in patients with rheumatoid arthritis. However, a significant proportion of patients does not achieve disease remission with methotrexate monotherapy, which can be attributed to multiple reasons. We hypothesize, that the efficacy limitations of this well-known medication can be, to some extent, overcome by sufficient dose and route optimisation. Furthermore, individual factors effecting the treatment response are unknown. Thus, we aim to evaluate the "maximised methotrexate therapy" before switching to biologic or targeted synthetic drugs.

The MethMax trial is a prospective, randomised, assessor-blinded, parallel-group, low-intervention trial, including 182 patients across 7 European countries. Patients with active rheumatoid arthritis, naïve to biologic or targeted synthetic antirheumatic drugs, who have been on a stable oral methotrexate therapy for the past 3 months will be randomised in 1:1 ratio to either 25mg oral or 25mg subcutaneous methotrexate weekly. In both arms, a short glucocorticoid therapy will be prescribed at baseline visit. The active study duration for each patient is 24 weeks. After inclusion, study visits take place at baseline, weeks 4, 8, 12, 16 and 24. The clinical efficacy and safety parameters will be obtained at each visit. At predefined timepoints, further patient reported outcomes, exploratory biomarkers like sweat and blood metabolites, as well as medication adherence will be assessed. Written consent will be obtained for all participants. The study has received regulatory approval via the Clinical Trials Information System and has recently started recruitment at the first centre.

The anticipated results will suggest whether the subcutaneous administration of 25mg methotrexate weekly is superior to oral methotrexate 25mg and lower doses in each route respectively. The outcomes include clinical disease activity, methotrexate metabolism analyses and medication adherence. The gained knowledge could lead to individual therapy optimisation and new therapy recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ≥ 18 years of age, capable of understanding and signing an informed consent (including sufficient literacy and proficiency in the local language) and following the study procedures
2. Patients with rheumatoid arthritis (RA) according to the 2010 American College of Rheumatology/European Alliance of Associations for Rheumatology (ACR/EULAR) classification criteria
3. Ongoing conventional therapy with oral methotrexate (between ≥10mg and 25mg weekly) for ≥3 months with stable dosing, and clinical and laboratory tolerance of this treatment for at least 12 weeks
4. CDAI > 2.8 + at least 1 clinically swollen joint (on 28-Joint count)
5. Willingness to increase methotrexate dosing and change the route of administration according to study procedures

Exclusion Criteria:

1. Inflammatory rheumatic diseases other than RA
2. Ongoing or previous therapy with any biological DiseaseModifying Anti-Rheumatic Drug (bDMARDs) or targeted synthetic DMARDs (tsDMARDs) or conventional synthetic DMARDs (csDMARDs) other than methotrexate and hydroxychloroquine
3. Use of GC unless on stable oral dose ≤10mg for at least 4 weeks prior to study inclusion
4. Patients using NSAIDs, unless taken at a stable dose for ≥2 weeks prior to study inclusion
5. Intraarticular GC treatment in the last 8 weeks
6. Patients with significant and clinically relevant MTX-drug toxicity as judged by the investigator
7. Elevated liver enzymes (aspartate transaminase (ASAT) and/or alanine transaminase (ALAT)), and/or alkaline phosphatase (AP), and/or gamma-glutamyl transferase (GGT) above 2x the upper limit normal (ULN)
8. Reduced kidney function (glomerular filtration rate (GFR)<60)
9. Haematologic abnormalities (grade 2 or 3: anaemia, leukopenia, thrombocytopenia)
10. Stomatitis under the treatment with MTX
11. Known history of recurrent/serious infections in the previous two months (such as, but not limited to, hepatitis, pneumonia, or pyelonephritis)
12. A positive HBsAg and/or HCV test at screening visit
13. Ongoing or recurring opportunistic infections (e.g., herpes zoster, cytomegalovirus, pneumocystis, aspergillosis, histoplasmosis, or mycobacteria) as judged by the investigator
14. Women of childbearing potential without the use of adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization) and willing to continue this precaution for the duration of the study until 6 months after receiving the last medication
15. Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, haematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease, as judged by the investigator
16. Being unable or unwilling to undergo multiple venepunctures because of poor tolerability or lack of sufficient venous access
17. Being unwilling or unable to perform s.c injections
18. Presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening)
19. Women who are pregnant, nursing; or planning pregnancy during the study and 6 months after the individual study completion
20. History of alcohol or substance abuse within the preceding 6 months
21. Any medical or psychological condition that, judged by the investigator, would interfere with safe completion of the trial
22. Immunisation with a live/attenuated vaccine within 12 weeks prior to baseline or potential need to receive a live vaccine during the course of the study
23. Active participation in any other interventional study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
CDAI remission (≤2.8) at week 24 | 24 weeks
  The primary endpoint is the achievement of remission defined as the CDAI ≤2.8 assessed 24 weeks after randomisation comparing patients with dose/route optimization (≥10mg MTX oral weekly switched to 25mg MTX subcutaneously weekly) and oral dose optimization (≥10mg MTX oral weekly switched to 25mg MTX oral weekly).

SECONDARY OUTCOMES:
CDAI low disease activity (≤10) at week 24 | 24 weeks
  To assess the proportion of patients in CDAI low disease activity (≤10) at week 24
CDAI remission (≤2.8) at week 12 | 12 weeks
  To assess the proportion of patients in CDAI remission (≤2.8) at week 12
CDAI low disease activity (≤10) at week 12 | 12 weeks
  To assess the proportion of patients in CDAI low disease activity (≤10) at week 12
ACR20% response at week 24 | 24 weeks
  To assess the proportion of patients achieving an ACR20% response at week 24
ACR20% response at week 12 | 12 weeks
  To assess the proportion of patients achieving an ACR20% response at week 12
ACR50% response at week 24 | 24 weeks
  To assess the proportion of patients achieving an ACR50% response at week 24
ACR50% response at week 12 | 12 weeks
  To assess the proportion of patients achieving an ACR50% response at week 12
ACR70% response at week 24 | 24 weeks
  To assess the proportion of patients achieving an ACR70% response at week 24
ACR70% response at week 12 | 12 weeks
  To assess the proportion of patients achieving an ACR70% response at week 12
Patient reported outcomes on NRS | 24 weeks
  Difference in change (absolute and relative) of patient reported outcomes on numeric response scale (NRS), including pain, patient global assessment, and joint stiffness between the treatment groups between baseline and week 24
Patient reported outcomes on NRS | 12 weeks
  Difference in change (absolute and relative) of patient reported outcomes on numeric response scale (NRS), including pain, patient global assessment, and joint stiffness between the treatment groups between baseline and week 24
Quality of Life questionnaires | 24 weeks
  Difference in change (absolute and relative) of patient reported outcomes measured by questionnaires:
  1. Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
  2. the 36-Item Short Form Survey version 1 (SF36v1)
  3. The Health Assessment Questionnaire Disability Index (HAQ-DI) between the treatment groups between baseline and week 12
Quality of Life questionnaires | 12 weeks
  Difference in change (absolute and relative) of patient reported outcomes measured by questionnaires:
  1. Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
  2. the 36-Item Short Form Survey version 1 (SF36v1)
  3. The Health Assessment Questionnaire Disability Index (HAQ-DI) between the treatment groups between baseline and week 12
Joint count and inflammatory markers | 24 weeks
  Difference in change (absolute and relative) of swollen joint count, tender joint count and CRP/ESR between baseline and week 24
Joint count and inflammatory markers | 12 weeks
  Difference in change (absolute and relative) of swollen joint count, tender joint count and CRP/ESR between baseline and week 12

OTHER OUTCOMES:
MTX-PGs levels and CDAI response | week 12 and 24
  Association of MTX-PGs levels and CDAI response at week 12 and week 24
Therapeutic drug monitoring (MTX metabolites, TTV) | week 12 and 24
  Association of MTX dosage, MTX-PGs levels and torque teno virus titer as a potential marker to guide levels of immunosuppressive therapy at week 12 and week 24
Finger sweat analysis | week 12 and 24
  Association of MTX-metabolites and inflammatory markers in finger sweat analysis and CDAI at week 12 and week 24
Cumulative glucocorticoid dose | 24 weeks
  Difference in cumulative glucocorticoid (GC) dose between treatment arms
Treatment adherence | 24 weeks
  Association of CDAI response and treatment adherence as measured by paper-based questionnaires, methotrexate metabolites and electronic adherence monitoring (in patients using the RheumaBuddy mobile app)
Safety profile | 24 weeks
  Differences in safety profile according to number of adverse events and organ systems (haematologic, hepatic, gastrointestinal, infections)
Trajectories of disease activity | 24 weeks
  Trajectories of disease activity in the two groups over all visits, and its relation to predictors

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
upon reasonable request